CLINICAL TRIAL: NCT02537028
Title: A Phase Ib Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Biological Effect of MSC2364447C in Systemic Lupus Erythematosus
Brief Title: MSC2364447C Phase 1b in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMR200527-002; 2015-001891-23 (EudraCT Number)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: MSC2364447C; Phase 1; BTK inhibitor; Systemic Lupus Erythematosus; M2951; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — evobrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSC2364447C 25 mg (Experimental)
  Interventions: Drug: MSC2364447C
- MSC2364447C 75 mg (Experimental)
  Interventions: Drug: MSC2364447C
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSC2364447C — Subjects will be administered with MSC2364447C 25 milligrams orally once daily for 4 weeks.
  Other Names: M2951, Evobrutinib
  Arms: MSC2364447C 25 mg
Drug: MSC2364447C — Subjects will be administered with MSC2364447C 75 milligrams orally once daily for 4 weeks.
  Other Names: M2951, Evobrutinib
  Arms: MSC2364447C 75 mg
Drug: Placebo — Subjects will be administered with placebo matching to MSC2364447C orally once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The primary purpose of this Phase 1b double-blind, randomized, placebo-controlled trial is to evaluate the safety, tolerability, pharmacokinetic (PK), and biological effect of MSC2364447C administered for 4 weeks in systemic lupus erythematosus subjects (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 to 65 years of age
* Diagnosis of systemic lupus erythematosus (SLE) (at least 4 of the 11 American College of Rheumatology [ACR] classification criteria for SLE) of at least 6 months duration at the Screening visit
* Positive test results for anti-nuclear antibody (ANA) (human epithelial cell-2 ANA greater than or equal to [>=] 1:80) and/or anti-dsDNA antibody (>= 30 international units per milliliter [IU/mL]) at the Screening visit
* At least 1 SLE disease manifestation (assessed by Systemic Lupus Erythematosus Disease Activity Index-2000 [SLEDAI-2K]) other than positive antidsDNA and no central nervous system (CNS) SLE (psychosis, organic brain syndrome, cranial nerve disorder, lupus headache, or new-onset cerebrovascular accident)
* History of vaccinations as follows or vaccination against these pathogens during Screening:

  1. Vaccination against Streptococcus pneumoniae with pneumococcal polysaccharide vaccine 23 or pneumococcal 13-valent conjugate vaccine as per local guidelines, and
  2. Vaccination against influenza virus (as per local seasonal recommendations). Subjects receiving 1 or more of these vaccinations during screening must have at least 2 weeks between the vaccination(s) and the date of randomization at Day 1.
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Active clinically significant CNS SLE
* Initiation or change in dose of anti-malarial treatment after the screening visit
* Within 2 weeks prior to Screening or during Screening: use of oral corticosteroids greater than (>) 40 mg daily prednisone equivalent, use of any injectable corticosteroids, or change in dose of corticosteroids
* Within 2 weeks prior to Screening, initiation or change in dose of angiotensin-converting enzyme inhibitor or angiotensin receptor blocker, or nonsteroidal anti-inflammatory drugs (NSAIDs).
* Within 2 months prior to Screening or during Screening: initiation of or change in dose of methotrexate, mycophenolate (mofetil or sodium), or azathioprine
* Within 2 months prior to Screening or during Screening, use of cyclosporine, tacrolimus, leflunomide, abatacept, anti-tumor necrosis factor alpha agents, intravenous immunoglobulin, plasmapheresis, or other disease-modifying, immunosuppressive, or immunomodulatory therapies not otherwise specified in protocol
* Within 6 months prior to Screening or during Screening: use of cyclophosphamide or chlorambucil
* Within 12 months prior to screening or during screening: use of rituximab, belimumab, or any other B cell-depleting or modulating therapies
* Within 1 month prior to Screening or during Screening, vaccination with live or live-attenuated virus vaccine.
* Active clinically significant viral, bacterial or fungal infection, or any serious episode of infection requiring hospitalization within the last 6 months - Estimated glomerular filtration rate by the Modification of Diet in Renal Disease equation of less than (<) 60 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2), or recent decline in kidney function, or proteinuria >= 3 gram per day (g/day) (spot urine protein/creatinine ratio >= 3 mg/mg)
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) | From the first dose of study drug administration up to 4 weeks after the last dose of study drug administration
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration up to 4 weeks after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.
Number of subjects with TEAEs according to severity | From the first dose of study drug administration up to 4 weeks after the last dose of study drug administration
  The severity of TEAEs will be graded using National cancer institute-Common Terminology Criteria for Adverse Events version 4.03 (NCI-CTCAE v 4.03) definitions of Grade 1 through Grade 5 following his/her best medical judgment. The severity of the AEs will be classified as follows: Grade 1 or mild, Grade 2 or moderate, Grade 3 or severe, Grade 4 or life-threatening and Grade 5 or death.
Number of subjects with clinically significant laboratory abnormalities | screening up to Day 56
  Clinical laboratory parameters being monitored for safety will be summarized using descriptive statistics, by postdose shifts relative to Baseline for relevant parameters using relevant cut-offs. Clinical significance will be determined by investigator.
Number of subjects with clinically significant abnormal vital signs: blood pressure, pulse rate, respiratory rate | screening up to Day 56
  Observed values and changes from Baseline in vital signs will be summarized for each treatment group using descriptive statistics. Clinically noteworthy changes in vital signs will be listed and summarized as appropriate. A semi-automated blood pressure and pulse rate recording device with an appropriate cuff size will be utilized. Blood pressure and pulse rate will be measured after 10 minutes' rest in the semi-supine position with the subject's arm unconstrained by clothing or other material. The blood pressure should be assessed on the same arm for each subject throughout the trial. Clinical significance will be determined by investigator.
Number of subjects with clinically significant abnormal electrocardiograms (ECGs) | screening up to Day 28
  Observed values and changes from Baseline in ECG will be summarized for each treatment group using descriptive statistics. Clinically noteworthy changes in ECG will be listed and summarized as appropriate. Clinical significance will be determined by investigator.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to 6 hours after administration (AUC0-6) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
Maximum observed plasma concentration (Cmax) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
Time to reach maximum plasma concentration (tmax) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
Concentration observed immediately before next dosing (Cpre) (Day 28) | Predose (within 30 minutes prior to dosing) on Day 28
Dose-normalized AUC0-6h (AUC0-6h/dose) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
Dose-normalized Cmax (Cmax/dose) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
Accumulation ratio for AUC0-6 (Racc(AUC0-6)) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
  Accumulation ratio for AUC will be calculated as AUC0-6, Day28 divided by AUC0-6, Day1
Accumulation ratio for Cmax (Racc(Cmax)) | Predose, 0.25, 0.5, 1.0, 2.0, 4.0, and 6.0 hours post-dose on Day 1 and Day 28
  Accumulation ratio for Cmax, calculated as Cmax, Day28 divided by Cmax, Day1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (11):
- United States (10):
  - Research site, Anniston, Alabama
  - Research site, El Cajon, California
  - Research site, Lakewood, California
  - Research site, Los Angeles, California
  - Research site, Clearwater, Florida
  - Research site, DeBary, Florida
  - Research site, Orlando, Florida
  - Research site, Grand Blanc, Michigan
  - Research site, St Louis, Missouri
  - Research site, Austin, Texas
- Research site, Sofia, Bulgaria